CLINICAL TRIAL: NCT03886220
Title: A Phase 4 Study to Evaluate the Safety and Efficacy of Elagolix for the Management of Heavy Menstrual Bleeding Associated With Uterine Fibroids in Premenopausal Women
Brief Title: A Study to Evaluate the Safety and Efficacy of Elagolix for the Management of Heavy Menstrual Bleeding Associated With Uterine Fibroids in Premenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-824
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Uterine Fibroids
Keywords: Elagolix; ABT-620; Uterine Fibroids; Heavy Menstrual Bleeding (HMB)
MeSH Terms: conditions — Leiomyoma; Menorrhagia | interventions — elagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Elagolix 150 mg (Experimental): Elagolix 150 mg once daily (QD)
  Interventions: Drug: Elagolix
- Placebo (Experimental): Placebo QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elagolix — Oral; Tablet
  Other Names: ABT-620; elagolix sodium; Orilissa
  Arms: Elagolix 150 mg
Drug: Placebo — Oral; Tablet
  Arms: Placebo

SUMMARY:
The main objective of this study is to assess safety and efficacy of elagolix compared to placebo in reducing heavy menstrual bleeding (HMB) associated with uterine fibroids in premenopausal women. The primary hypothesis is that elagolix, compared to placebo, reduces HMB associated with uterine fibroids in premenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Participant at the time of screening has a diagnosis of uterine fibroids documented by a pelvic ultrasound [transabdominal ultrasound (TAU) and transvaginal ultrasound (TVU)].
* Participant has HMB associated with uterine fibroids as evidenced by menstrual blood loss (MBL) > 80 mL during 1 menses in screening as measured by the alkaline hematin method.
* Participant has negative urine and/or serum pregnancy test in Washout (if applicable) and/or Screening and just prior to first dose.
* Participant has an adequate endometrial biopsy performed during Screening, the results of which show no clinical significant endometrial pathology.

Exclusion Criteria:

* Participant has screening pelvic ultrasound or saline infusion sonohysterography (SIS) or magnetic resonance imaging (MRI; if SIS is unevaluable), results that show a clinically significant gynecological disorder.
* Participant has history of osteoporosis, osteopenia, or other metabolic bone disease.
* Participant has clinically significant abnormalities in clinical chemistry, hematology, or urinalysis.
* Participant has a history of major depression or post-traumatic stress disorder (PTSD) episode within 2 years of screening, OR a history of other major psychiatric disorder at any time (e.g., schizophrenia, bipolar disorder).
* Participant is using any systemic corticosteroids for over 14 days within 3 months prior to Screening or is likely to require treatment with systemic corticosteroids during the course of the study. Over the counter and prescription topical, inhaled, intranasal or intra-articular injectable (for occasional use) corticosteroids are allowed.

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (48):
- United States (45):
  - ACCEL Research Sites /ID# 209714, Birmingham, Alabama
  - University of Alabama at Birmingham - Women's and Infant's Center /ID# 209581, Birmingham, Alabama
  - Unity Health- Searcy Medical Center /ID# 210905, Searcy, Arkansas
  - Grossmont Ctr Clin Research /ID# 217690, La Mesa, California
  - Women's Health Care Research Corp /ID# 211472, San Diego, California
  - Alliance for Multispecialty Research (AMR) - Fort Myers /ID# 213764, Fort Myers, Florida
  - Caceres Specialized Gynecology /ID# 214956, Kissimmee, Florida
  - LCC Medical Research Institute /ID# 213765, Miami, Florida
  - Genoma Research Group, Inc /ID# 213771, Miami, Florida
  - A Premier Medical Research of FL /ID# 214947, Orange City, Florida
  - GCP Clinical Research, LLC /ID# 218742, Tampa, Florida
  - Comprehensive Clinical Trials LLC /ID# 217177, West Palm Beach, Florida
  - Georgia Research for Women /ID# 211321, Atlanta, Georgia
  - Atlanta Women's Research Institute /ID# 217745, Atlanta, Georgia
  - Medisense Inc /ID# 217750, Atlanta, Georgia
  - Women's Health of Augusta /ID# 214995, Augusta, Georgia
  - Midtown OBGYN North /ID# 209391, Columbus, Georgia
  - Journey Medical Research Institute - Snellville /ID# 217309, Snellville, Georgia
  - Affinity Clinical Research /ID# 215252, Oak Brook, Illinois
  - Clinical Trials Management, LLC - Covington /ID# 215020, Covington, Louisiana
  - Southern Clinical Research A /ID# 213732, Metairie, Louisiana
  - Johns Hopkins University /ID# 211135, Baltimore, Maryland
  - NECCR Fall River LLC /ID# 215009, Fall River, Massachusetts
  - Excel Clinical Research /ID# 215936, Las Vegas, Nevada
  - Manhattan Medical Research /ID# 213753, New York, New York
  - Upstate Clinical Research Associates /ID# 215156, Williamsville, New York
  - M3 Wake Research Inc. /ID# 215166, Raleigh, North Carolina
  - Carolina Medical Trials - Winston-Salem /ID# 215027, Winston-Salem, North Carolina
  - Legacy Medical Group-Gynecologic Oncology /ID# 211016, Portland, Oregon
  - Clinical Research of Philadelphia, LLC /ID# 213741, Philadelphia, Pennsylvania
  - Reading Hospital Clinical Trials Office /ID# 213763, West Reading, Pennsylvania
  - Clinical Trials of SC /ID# 210204, Charleston, South Carolina
  - Chattanooga Medical Research /ID# 215294, Chattanooga, Tennessee
  - WR-Medical Research Center of Memphis LLC /ID# 213756, Memphis, Tennessee
  - Access Clinical Trials, Inc. /ID# 215357, Nashville, Tennessee
  - Signature Gyn Services /ID# 213883, Fort Worth, Texas
  - FMC Science, LLC - OB/GYN - Georgetown /ID# 211164, Georgetown, Texas
  - University of Texas (UT) Health Women's Research Center at Memorial City /ID# 215193, Houston, Texas
  - Advances in Health, Inc. /ID# 215847, Houston, Texas
  - Clinical Trials of Texas, Inc /ID# 213768, San Antonio, Texas
  - Discovery Clinical Trials-San Antonio /ID# 214996, San Antonio, Texas
  - Storks Research, LLC /ID# 211146, Sugar Land, Texas
  - Houston Ctr for Clin Research /ID# 215138, Sugar Land, Texas
  - Seattle Clinical Research Center /ID# 210853, Seattle, Washington
  - North Spokane Women's Health /ID# 209889, Spokane, Washington
- Puerto Rico (3):
  - Emanuelli Research & Development Center LLC /ID# 212715, Arecibo
  - Puerto Rico Medical Research /ID# 212841, Ponce
  - Mindful Medical Research /ID# 212496, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Brown E, Kroll R, Li H, Ng J, Pinsky B, Rodriguez JW, Thomas J, Snabes MC. Low-Dose Elagolix for the Treatment of Heavy Menstrual Bleeding in Patients With Uterine Leiomyomas: A Randomized Controlled Trial. Obstet Gynecol. 2023 Nov 1;142(5):1068-1076. doi: 10.1097/AOG.0000000000005380. Epub 2023 Sep 28. PMID 37769311
- See also: Related Info — https://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo once daily (QD)
- Elagolix 150 mg: Elagolix 150 mg QD
Period: Treatment Period
Arm/Group | Placebo | Elagolix 150 mg
Started | 28 | 54
Completed (Completed study drug treatment.) | 23 | 42
Not Completed | 5 | 12
Not completed — Discontinued study drug during the treatment period | 5 | 12
Period: Post-Treatment Follow-Up Period
Arm/Group | Placebo | Elagolix 150 mg
Started (Entered the post-treatment follow-up period (includes some participants who discontinued study drug during the treatment period).) | 25 | 41
Completed | 23 | 39
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Elagolix 150 mg | Total
Number analyzed (Participants) | 28 | 54 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (3.82) | 42.0 (5.02) | 42.3 (4.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 54 | 82
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 12 | 18
  Not Hispanic or Latino | 22 | 42 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 16 | 27
  Black or African American | 17 | 37 | 54
  Asian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Responders With Menstrual Blood Loss (MBL) Volume < 80 mL at Final Month and >= 50% Reduction in MBL Volume From Baseline to the Final Month
Description: Responders were defined as participants meeting the following 2 conditions:
  * menstrual blood loss (MBL) volume < 80 mL at the Final Month (defined as the last 28 days prior to and including the last dose day), and
  * 50% or greater reduction in MBL volume from Baseline to the Final Month.
  Participants whose primary reason for prematurely discontinuing study drug was "lack of efficacy," or "requires surgery or invasive intervention for treatment of uterine fibroids" were considered as non-responders. MBL was measured by the alkaline hematin method.
Time Frame: From Month 0 (Baseline) to Final Month (up to Month 6)
Population: Full Analysis Set; multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 28 | 54
percentage of participants | 23.3 [7.16 to 39.50] | 49.4 [35.06 to 63.83]
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Test type: Superiority; p = 0.035, Regression, Logistic — P-value for test of difference between elagolix dose group and placebo is by pooling the results from a logistic regression model including treatment as the main effect and baseline MBL volume as a covariate in each dataset from multiple imputation; Odds Ratio (OR) = 3.22, 95% CI 2-sided [1.086 to 9.546]

ADVERSE EVENTS:
Time Frame: All-cause mortality: median of 197 days. Serious adverse events/other adverse events: from first dose of study drug through Month 7.
Arm/Group | Placebo | Elagolix 150 mg
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/54
Serious Adverse Events (participants affected / at risk) | 2/28 | 0/54
Other Adverse Events (participants affected / at risk) | 2/28 | 11/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Elagolix 150 mg (N=54)
ENLARGED UVULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Elagolix 150 mg (N=54)
HEADACHE (Nervous system disorders) | 1 (1) | 7 (7)
HOT FLUSH (Vascular disorders) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT03886220/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT03886220/SAP_001.pdf